CLINICAL TRIAL: NCT02086994
Title: Carbetocin in Preventing Postpartum Bleeding in Women With Severe Preeclampsia.
Brief Title: Prevention of Postpartum Hemorrhage in Patients With Severe Preeclampsia Using Carbetocin Versus Misoprostol
Acronym: carbetocin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: khalid abd aziz mohamed (Other)
Responsible Party: Sponsor-Investigator, khalid abd aziz mohamed, lecturer, Benha University
Organization: Benha University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: khalid77
Record Dates: First submitted 2014-03-05; First posted 2014-03-14 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Severe Pre-eclampsia, Postpartum Condition or Complication
Keywords: carbetocin, misoprostol, pre-eclampsia, pph
MeSH Terms: conditions — Pre-Eclampsia; Familial Primary Pulmonary Hypertension | interventions — Misoprostol; carbetocin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cabetocin (Active Comparator): a single dose of carbetocin (100 μg in 1 mL ampoule, Pabal) given intravenously after delivery of anterior shoulder
  Interventions: Drug: carbetocin
- misoprostol (Active Comparator): misoprostol (600 μg, 3 tables) sublingually after the delivery of the anterior shoulder of the baby.
  Interventions: Drug: misoprostol

INTERVENTIONS:
Drug: misoprostol — given after the delivery of the anterior shoulder of the baby.
  Other Names: misoprost; cytotec; misotec
  Arms: misoprostol
Drug: carbetocin — given after delivery of anterior shoulder
  Other Names: pabal
  Arms: cabetocin

SUMMARY:
We aim to compare carbetocin with misoprostol for the prevention of postpartum hemorrhage in patients with severe preeclampsia. The primary outcome is postpartum haemorrhage (blood loss of ≥ 500 ml) while our Secondary outcomes include use of additional uterotonics, need for blood transfusion, maternal adverse drug reaction, maternal complications and maternal death

DETAILED DESCRIPTION:
We conducted a prospective non-randomized study at Department of Obstetrics and Gynecology, Benha University Hospital, since March 2013 till June 2015, after approval of the study protocol by the Local Ethical Committee. A written informed consent was obtained from eligible women before induction or at early stage of labour.

Women with singleton pregnancies of more than 28 weeks' gestation who are admitted to hospital with severe preeclampsia and candidates for vaginal delivery were eligible for the study. Preeclampsia is labelled as severe in the presence of any of the following abnormalities.

1. Persistent cerebral or visual disturbances or cerebral edema.
2. Persistent epigastric pain with nausea or vomiting, or both.
3. Systolic ≥160 mmHg or diastolic ≥110 mmHg on 2 occasions at least 6 h apart with the patient at bed rest.
4. Proteinuria of ≥5 g on 24-hour urine collection. Urine dipsticks are not accurate for this purpose.
5. Oliguria (˂500 mL in 24 hours).
6. Pulmonary edema.
7. Thrombocytopenia.

Our exclusion criteria are HELLP syndrome, eclampsia, abruptio placentae, malpresentation, polyhydramnios, previous uterine scar, chorioamnionitis and multiple pregnancies. All patients were in stable condition (no evidence of maternal hemodynamic instability or fetal distress) and their management afterwards followed the standards accepted in our country and established guidelines for the management of hypertensive disorders of pregnancy. For hypertensive crisis the first drug used was hydralazine (5 mg IV every 15 minutes to a maximum total dose of 20 mg) and, if this was ineffective, Nifedipine (Epilat): 10 to 20 mg orally / 30 min (max 50 mg), Then 10-20 mg /4-6 h (max 120 mg/day) or labetalol (20 mg IV every 10 minutes to a maximum total dose of 300 mg). No patient needed additional treatment for their symptoms or developed antepartum complications that required admission to the intensive care unit. All patients were evaluated hourly and received magnesium sulphate to prevent eclampsia during the pregnancy and for a minimum of 24 hours postpartum.

The patients (60) were divided into two groups, Group A (30) received a single dose of carbetocin (100 μg in 1 mL ampoule, Pabal) while Group B (30) received misoprostol (600 μg, 3 tables) sublingually after the delivery of the anterior shoulder of the baby.

The third stage of labour is managed as usual by clamping and cutting of umbilical cord, waiting for signs of placental separation and delivering the placenta by controlled cord traction.

Duration of the 3rd stage of labour is calculated. Patient is kept in labor room under observation for a period of 1 h and any complaint such as nausea, vomiting, fever, headache, chills, diarrhoea and shivering is noted. In cases of uterine atony (determined by physical examination and continuous postpartum bleeding) uterus is massaged and additional uterotonics were given and noted (oxytocin and/or prostaglandin, at the discretion of the attending physician). Any requirement for manual removal of the placenta or blood transfusion is also recorded.

The following laboratory assessments (hemoglobin, hematocrit, platelets, and renal and liver function tests) are performed in every patient on admission and postpartum. Vital signs (blood pressure, heart rate, respiratory rate) and urine output are measured every hour until at least 24 hours after delivery.

Measurement of blood loss A clean plastic lined absorbent drape is placed under the woman's buttocks to collect all the blood lost after delivery of the baby and drainage of the amniotic fluid. The drape is changed as many times as needed. The woman stays on the drape or asked to wear a pad over the next 60 minutes. In the case of severe haemorrhage, we follow the usual guidelines for management of postpartum haemorrhage, and the supplemental treatment is registered. All drapes and pads are weighed on an electronic scale and the known dry weight of the linen is subtracted. As 1 ml of blood weighs close to 1 g, the balance in grams is assumed to be the total blood loss in ml.

Haemoglobin concentration is measured before, 2 hours and 24 hours after delivery.

The rate of haemorrhage at labour third phase is determined by observation estimation considering the amount of blood under the patient. The rate of haemoglobin and haematocrit are measured at hospitalization and also 2 h, 24 h after delivery and then are recorded. At this interval, the patients are evaluated in terms of possible complications of administered drugs such as vomiting, diarrhoea, shivering, pyrexia, and headache).

All patients have the Foley catheter in situ for 24 hours after delivery and the amount of urine was monitored hourly.

This study has no external funding source. No author had any potential relationships that may pose conflict of interest.

Outcome measures Our primary outcome measure is postpartum haemorrhage, defined as a blood loss of ≥ 500 ml. We analyse the blood loss, change in haemoglobin concentration between admission and discharge. While secondary outcomes include use of additional uterotonics, need for blood transfusion, maternal adverse drug reaction (such as headache, vomiting, abdominal pain, pruritus, tacky or bradycardia), sever maternal complications (such as seizures or need for ICU admission) and maternal death.

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton pregnancies of more than 28 weeks' gestation who were admitted to hospital with severe preeclampsia and candidates for vaginal delivery were eligible for the study. Preeclampsia is labelled as severe in the presence of any of the following abnormalities:

  1. Persistent cerebral or visual disturbances or cerebral edema.
  2. Persistent epigastric pain with nausea or vomiting, or both.
  3. Systolic ≥160 mmHg or diastolic ≥110 mmHg on 2 occasions at least 6 h apart with the patient at bed rest.
  4. Proteinuria of ≥5 g on 24-hour urine collection. Urine dipsticks are not accurate for this purpose.
  5. Oliguria (˂500 mL in 24 hours).
  6. Pulmonary edema.
  7. Thrombocytopenia.

Exclusion Criteria:

* were HELLP syndrome, eclampsia, abruptio placentae, malpresentation, polyhydramnios, previous uterine scar, chorioamnionitis and multiple pregnancies

Ages: 19 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Prevention of postpartum hemorrhage in patients with severe preeclampsia using carbetocin versus misoprostol | 24 hours after delivery
  prevention of postpartum haemorrhage

SECONDARY OUTCOMES:
measurement of blood loss during second stage of labour | 24 hours after delivery

CONTACTS AND LOCATIONS:
Overall Officials: khalid mohamed, MD, Study Chair — lecturer of ob/gyn Benha faculty of medicine; ahmed sasd, MD, Principal Investigator — lecturer; ahmed walid, Principal Investigator — assistant profossor
Locations (1):
- Benha univesity hospital, Banhā, Egypt